CLINICAL TRIAL: NCT02742259
Title: Prospective, Multi-Center Validation of the Prostate Cancer Assay
Brief Title: Validation of the Prostate Cancer Assay - Beta+Pivotal
Acronym: VPCA-B+PIV
Status: Withdrawn | Type: Observational
Why Stopped: No enrolled participants
Sponsor: Celsee Diagnostics (Industry)
Responsible Party: Sponsor
Other Study IDs: Celsee CA1001.v1
Record Dates: First submitted 2016-03-24; First posted 2016-04-19 (Estimated); Last update posted 2019-03-26 (Actual); Status verified 2019-03

CONDITIONS: Metastatic Prostate Cancer, CTC
MeSH Terms: conditions — Prostatic Neoplasms; Neoplastic Cells, Circulating | interventions — Blood Specimen Collection

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: None Retained — 10 ml blood draws
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

GROUPS / COHORTS (2):
- Beta Cutoff: Assay
  Interventions: Device: Blood Draw
- Pivotal: Assay
  Interventions: Device: Blood Draw

INTERVENTIONS:
Device: Blood Draw — Blood draws only - non-diagnostic, non-treatment

SUMMARY:
The Prostate Cancer Assay performance of Celsee Diagnostics circulating tumor cell (CTC) analysis system will be validated in patients diagnosed with metastatic prostate cancer. It will demonstrate substantial performance equivalency to a CTC Assay predicate device.

ELIGIBILITY:
Inclusion Criteria:

* • Male aged 18 years and above

  * Be willing to sign an informed consent document indicating that the subject understands the purpose of and procedures required for the study and are willing to participate in the study
  * Be willing/able to adhere to the prohibitions and restrictions specified in this protocol
  * Eastern cooperative group (ECOG) performance status ≤2
  * Documented histologically confirmed adenocarcinoma of the prostate
  * Metastatic prostate cancer to the bone as documented by positive bone scan imaging
  * CRPC patient being considered for systemic therapy or in between lines of therapies (>= 14 days from prior treatment) for metastatic disease. Patient must have evidence of castrate resistant prostate cancer as evidenced by a confirmed rising PSA (per Prostate Cancer Working Group 2 [PCWG2] criteria) and a castrate serum testosterone level (i.e. ≤ 50 mg/dl).

Exclusion Criteria:

* • Subjects actively receiving systemic therapy regimens, or between lines of therapies (< 14 days from prior treatment)

  * Have any condition that, in the opinion of the investigator, would compromise the wellbeing of the subject or the study or prevent the subject from meeting or performing study requirements
  * Active infection or other medical condition that would make corticosteroids (i.e. prednisone) use contraindicated
  * Uncontrolled hypertension (systolic BP ≥ 160 mmHg or diastolic BP ≥ 95 mmHg) Patients with a history of hypertension are allowed provided blood pressure is controlled by antihypertensive treatment
  * Severe hepatic impairment (Child-Pugh Class C)
  * History of pituitary or adrenal dysfunction (note: the use of daily steroids does not exclude someone from participating in this study)
  * Have poorly controlled diabetes (HgB A1C ≥ 8%)
  * Any psychological, familial, sociological, or geographical condition that could potentially interfere with compliance with the study protocol and follow-up schedule.
  * Abnormal bone marrow function (absolute neutrophil count [ANC] < 1500/mm3, platelet count <100,000/mm3, hemoglobin <9 g/dL)
  * Abnormal liver function (bilirubin > upper limit of normal [ULN]; AST and/or ALT > 1.5 x ULN concomitant with alkaline phosphatase > 2.5 x ULN)
  * Abnormal kidney function (serum creatinine ≥ 2 x upper limit of normal)
  * Clinically significant heart disease as evidenced by myocardial infarction, or arterial thrombotic events in the past 6 months, severe or unstable angina, unstable atrial fibrillation, or New York Heart Association (NYHA) Class III-IV heart disease
  * History of ventricular tachyarrhythmia within the past 5 years

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Males 18 years and above; Metastatic prostate cancer to the bone as documented by positive bone scan imaging
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2016-05 (Estimated); Primary Completion 2017-04 (Estimated); Study Completion 2017-09 (Estimated)

PRIMARY OUTCOMES:
Confirmation of the clinical utility of the cutoff level for the Prostate Cancer Assay for prognosis of progression free survival (PFS) in comparison to the predicate device, CellSearch CTC Assay | 9 months
  "CTC negative" means a level of CTCs below the cutoff indicating lower risk for progression (i.e. PFS, and "CTC positive" means a level of CTCs at or above the cutoff indicating higher risk for progression (i.e. shorter PFS).

CONTACTS AND LOCATIONS:
Overall Officials: Yixin Wang, Ph.D., Study Director — Celsee Diagnostics

IPD SHARING:
Plan to Share IPD: No